CLINICAL TRIAL: NCT06747208
Title: The Impact of Swallowing and Nutrition in Head and Neck Cancer Patients Undergoing Chemo or Chemo-radiotherapy.
Brief Title: Dysphagia in Head and Neck Cancer With Radiation
Status: Not yet recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Clinical Trial Center, Attending Anesthesiologist, National Taiwan University Hospital
Other Study IDs: 202410077DINE
Record Dates: First submitted 2024-12-15; First posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Swallowing Function
Keywords: dysphagia; head and neck cancer; radiation therapy
MeSH Terms: conditions — Deglutition Disorders; Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — the DNA associated with nutrition
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- head and neck cancer patients: patients with head and neck cancer undergoing radiation therapy

SUMMARY:
This study focuses on swallowing dysfunction, a common issue affecting 60-75% of head and neck cancer patients due to tumor damage, treatment complications, and chemoradiotherapy side effects, which can lead to malnutrition and reduced quality of life. With limited research on the effects of radiation doses on swallowing muscles and nutrition, this study aims to evaluate these impacts in non-surgical patients undergoing radiotherapy, conducting assessments before treatment, three months after, and within one year post-treatment.

DETAILED DESCRIPTION:
Swallowing dysfunction is a common and debilitating symptom in head and neck cancer patients, affecting approximately 60-75% during the disease course, primarily due to tumor destruction, postoperative complications, and side effects of radiotherapy and chemotherapy. Combined chemoradiotherapy exacerbates adverse effects, such as mucositis, odynophagia, taste alterations, xerostomia, nausea, vomiting, and fatigue, which can result in dehydration, significant weight loss, and detrimental impacts on nutritional status, functionality, and quality of life. Limited research exists on the effects of radiation and chemoradiation doses on swallowing muscles, quality of life, and nutritional changes in these patients. This study aims to evaluate the impact of radiation doses on swallowing muscles and quality of life in head and neck cancer patients undergoing chemoradiotherapy while identifying malnutrition risk in this population. Non-surgical patients receiving radiotherapy as the primary treatment will be recruited, with swallowing, muscle, and nutritional assessments conducted before treatment, three months after treatment, and within one year post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo radiotherapy or concurrent chemoradiotherapy ;
* Aged between 18 and 80 years;
* Able to perform self-care independently (ECOG ≤ 2);
* All patients provide written informed consent.

Exclusion Criteria:

* Patients scheduled to undergo surgical treatment;
* Patients with neuromuscular diseases, such as stroke or Parkinson's disease;
* Patients with other diseases or complications, including heart disease classified as NYHA functional class ≥ 2 with thrombotic conditions, or lung disease classified as Hugh-Jones grade ≥ 4;
* Patients with psychological disorders that may affect their ability to provide informed consent or comply with the study protocol;
* Patients who do not consent to undergo high-resolution impedance manometry.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with head and neck cancer undergoing radiation therapy
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
hypopharyngeal mean peak pressure | one year
  hypopharyngeal contraction

IPD SHARING:
Plan to Share IPD: No
due to ethical issue